CLINICAL TRIAL: NCT00084266
Title: Linezolid In The Treatment Of Subjects With Nosocomial Pneumonia Proven To Be Due To Methicillin-Resistant Staphylococcus Aureus
Brief Title: Nosocomial Pneumonia With Suspected Or Proven Methicillin-Resistant Staphylococcus Aureus (MRSA)
Acronym: ZEPHYR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A5951001
Record Dates: First submitted 2004-06-09; First posted 2004-06-11 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Methicillin Resistant Staphylococcus Aureus (MRSA)
Keywords: Staphylococcal pneumonia; Methicillin-resistant staphylococcal pneumonia; healthcare-associated pneumonia
MeSH Terms: conditions — Pneumonia, Staphylococcal; Healthcare-Associated Pneumonia | interventions — Linezolid; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects receiving linezolid for the treatment phase of the study
  Interventions: Drug: linezolid (Zyvox)
- 2 (Active Comparator): Subjects receiving vancomycin for the treatment phase of the study
  Interventions: Drug: vancomycin

INTERVENTIONS:
Drug: linezolid (Zyvox) — Subjects to receive either linezolid 600 mg IV (Intravenous) or PO (orally) q 12 h (every 12 hours) for 7-14 days, except in cases of documented bacteremia where it could be extended to 21 days based upon investigator's discretion.
  Other Names: Zyvox, linezolid
  Arms: 1
Drug: vancomycin — Subjects to receive vancomycin 15mg/kg IV (Intravenous) q12h (every 12 hours), adjusted for renal function, for 7-14 days, except in cases of documented bacteremia where it could be extended to 21 days based upon investigator's discretion.
  Arms: 2

SUMMARY:
To determine if linezolid is superior to vancomycin in the treatment of nosocomial (acquired in the hospital) pneumonia due to Methicillin Resistant Staphylococcus Aureus (MRSA) in adult subjects. Subjects entered in to the study will have proven healthcare-associated methicillin-resistant Staphylococcus aureus pneumonia which will be treated with either linezolid or vancomycin.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male and female subjects with clinically documented nosocomial pneumonia proven to be due to methicillin-resistant staphylococcus aureus.
* Chest X-ray at baseline/screen or within 48 hours of treatment consistent with the diagnosis of pneumonia.
* Suitable sputum specimen defined as having less than 10 squamous epithelial cells and greater or equal 25 leukocytes or have a culture taken by an invasive technique within 24 hours of study entry.

Exclusion Criteria:

* Subjects who were treated with a previous antibiotic with MRSA activity (other than linezolid or vancomycin) for more than 48 hours, unless documented to be a treatment failure (72 hours of treatment and not responding).
* Subjects with severe neutropenia (<500 cells/mm3)
* Subjects with hypersensitivity to oxazolidinones or vancomycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1225 (Actual)
Dates: Start 2004-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (131):
- United States (74):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Redlands, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Brandon, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Jackson, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, North Chicago, Illinois
  - Pfizer Investigational Site, Oak Park, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, New Albany, Indiana
  - Pfizer Investigational Site, Hazard, Kentucky
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Saint Loius, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Reno, Nevada
  - Pfizer Investigational Site, Hackensack, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Greensboro, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Sylvania, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Abington, Pennsylvania
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Sioux Falls, South Dakota
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, San Marcos, Texas
  - Pfizer Investigational Site, Sequin, Texas
  - Pfizer Investigational Site, Temple, Texas
  - Pfizer Investigational Site, Murray, Utah
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Winchester, Virginia
- Pfizer Investigational Site, Buenos Aires, Buenos Aires, Argentina
- Belgium (4):
  - Pfizer Investigational Site, Bruges
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Liège
- Brazil (3):
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, São José do Rio Preto, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Chile (3):
  - Pfizer Investigational Site, Santiago, RM
  - Pfizer Investigational Site, Santiago, Santiago Metropolitan
  - Pfizer Investigational Site, Santiago
- Colombia (4):
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogotá, Bogota. DC
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Ibagué, Tolima Department
- France (4):
  - Pfizer Investigational Site, Paris, Cedex 18
  - Pfizer Investigational Site, Marseille, France
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Saint-Etienne
- Germany (2):
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Leipzig
- Greece (4):
  - Pfizer Investigational Site, Kifissia, Athens
  - Pfizer Investigational Site, Crete, Greece
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Thessaloniki
- Pfizer Investigational Site, Hong Kong, Hong Kong
- Pfizer Investigational Site, Kuala Lumpur, Malaysia
- Mexico (4):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Monterrey/Col. Mitras Centro, Nuevo Léon
  - Pfizer Investigational Site, Ciudad Madero, Tamaulipas
- Poland (3):
  - Pfizer Investigational Site, Bytom
  - Pfizer Investigational Site, Katowice
  - Pfizer Investigational Site, Krakow
- Portugal (4):
  - Pfizer Investigational Site, Almada
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Senhora da Hora
- Puerto Rico (2):
  - Pfizer Investigational Site, Ponce
  - Pfizer Investigational Site, San Juan
- Russia (2):
  - Pfizer Investigational Site, Moscow, Russia
  - Pfizer Investigational Site, Moscow
- South Africa (3):
  - Pfizer Investigational Site, Auckland Park
  - Pfizer Investigational Site, Bloefontein
  - Pfizer Investigational Site, Soweto
- Pfizer Investigational Site, Seoul, South Korea
- Spain (3):
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
- Taiwan (4):
  - Pfizer Investigational Site, Banqiao District
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
- Pfizer Investigational Site, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - Pfizer Investigational Site, Plymouth, Devon
  - Pfizer Investigational Site, Edinburgh
- Pfizer Investigational Site

REFERENCES:
- [Derived] Equils O, da Costa C, Wible M, Lipsky BA. The effect of diabetes mellitus on outcomes of patients with nosocomial pneumonia caused by methicillin-resistant Staphylococcus aureus: data from a prospective double-blind clinical trial comparing treatment with linezolid versus vancomycin. BMC Infect Dis. 2016 Sep 6;16(1):476. doi: 10.1186/s12879-016-1779-5. PMID 27600290
- [Derived] Shorr AF, Puzniak LA, Biswas P, Niederman MS. Predictors of Clinical Success in the Treatment of Patients with Methicillin-Resistant Staphylococcus aureus (MRSA) Nosocomial Pneumonia (NP). PLoS One. 2015 Jul 21;10(7):e0131932. doi: 10.1371/journal.pone.0131932. eCollection 2015. PMID 26196695
- [Derived] Quartin AA, Scerpella EG, Puttagunta S, Kett DH. A comparison of microbiology and demographics among patients with healthcare-associated, hospital-acquired, and ventilator-associated pneumonia: a retrospective analysis of 1184 patients from a large, international study. BMC Infect Dis. 2013 Nov 27;13:561. doi: 10.1186/1471-2334-13-561. PMID 24279701
- [Derived] Puzniak LA, Morrow LE, Huang DB, Barreto JN. Impact of weight on treatment efficacy and safety in complicated skin and skin structure infections and nosocomial pneumonia caused by methicillin-resistant Staphylococcus aureus. Clin Ther. 2013 Oct;35(10):1557-70. doi: 10.1016/j.clinthera.2013.08.001. Epub 2013 Sep 3. PMID 24011955

RESULTS

PARTICIPANT FLOW:
Groups:
- Linezolid: Linezolid intravenous (IV) approximately every 12 hours (twice daily) at a dose of 600 milligrams (mg) infused over a period of 60-120 minutes for 7 to 14 days except in cases of documented bacteremia where it could be extended to 21 days based upon investigator's discretion.
- Vancomycin: Vancomycin IV approximately every 12 hours (twice daily) at a dose of 30 mg/kg/day in 2 divided doses (15 mg/kg/dose) over a period of 60-120 minutes for 7 to 14 days except in cases of documented bacteremia where it could be extended to 21 days based upon investigator's discretion.
Period: Overall Study
Arm/Group | Linezolid | Vancomycin
Started | 618 | 607
Treated | 597 | 587
Completed | 177 | 184
Not Completed | 441 | 423
Not completed — Death | 42 | 39
Not completed — Adverse Event | 8 | 5
Not completed — Lack of Efficacy | 2 | 4
Not completed — Lost to Follow-up | 5 | 3
Not completed — Participant not willing to participate | 3 | 8
Not completed — Other | 360 | 344
Not completed — Randomized not treated | 21 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Linezolid | Vancomycin | Total
Number analyzed (Participants) | 597 | 587 | 1184
Age Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (18.4) | 60.5 (18.4) | 60.5 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 207 | 409
  Male | 395 | 380 | 775
Clinical Signs and Symptoms for modified intent-to-treat (mITT) Population [Number; unit: Participants] — Clinical signs and symptoms (mild to severe):cough;production of purulent sputum;auscultatory finding on pulmonary examination of rales,pulmonary consolidation(dullness on percussion, bronchial breath sounds,egophony);dyspnea, tachypnea,hypoxemia with partial pressure of oxygen(PaO2)<60 mmHg/worsening gas exchange/increased O2 requirement.
  Participants
    Decreased Breath Sounds | 169 | 182 | 351
    Hypoxia | 164 | 151 | 315
    Pulmonary Consolidation | 173 | 184 | 357
    Rales | 172 | 177 | 349
    Tachypnea | 152 | 143 | 295
    Chills/Rigors | 22 | 11 | 33
    Cough | 122 | 107 | 229
    Dyspnea | 99 | 95 | 194
    Pleuritic Chest Pain | 14 | 12 | 26
    Purulent Sputum | 167 | 209 | 376
Clinical Signs and Symptoms for Per Protocol (PP) Population [Number; unit: Participants] — Clinical signs and symptoms (mild to severe):cough;production of purulent sputum;auscultatory finding on pulmonary examination of rales,pulmonary consolidation(dullness on percussion, bronchial breath sounds,egophony);dyspnea, tachypnea,hypoxemia with PaO2<60 mmHg/worsening gas exchange/increased O2 requirement.
  Participants
    Decreased Breath Sounds | 138 | 155 | 293
    Hypoxia | 133 | 127 | 260
    Pulmonary Consolidation | 145 | 158 | 303
    Rales | 142 | 149 | 291
    Tachypnea | 124 | 123 | 247
    Chills/Rigors | 18 | 9 | 27
    Cough | 101 | 90 | 191
    Dyspnea | 80 | 80 | 160
    Pleuritic Chest Pain | 12 | 9 | 21
    Purulent Sputum | 171 | 174 | 345

OUTCOME MEASURES:

1. Primary Outcome: Clinical Outcome in Participants With Baseline Methicillin Resistant Staphylococcus Aureus (MRSA) at End of Study (EOS) for PP Population
Description: Clinical response was based primarily on global assessment of clinical presentation of participant made by investigator at evaluation timepoint. Clinical response was evaluated at EOS Visit as Cure: resolution of clinical signs/symptoms of pneumonia when compared with baseline; Failure: persistence/progression of baseline signs/symptoms of pneumonia or baseline radiographic abnormalities after atleast 2 days of treatment; development of new pulmonary/extrapulmonary clinical findings consistent with active infection; Unknown:extenuating circumstances precluding classification to 1 of the above.
Time Frame: EOS (7-30 days after last dose)
Population: PP population included all mITT participants who satisfied all critical inclusion/exclusion criteria,had adequate dosing of drug (defined as 5 full days for success or 2 full days of treatment for participants whose clinical outcome was considered failure) and had observed outcome for that visit unless already declared failure prior to that visit.
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 165 | 174
Participants
  Cure | 95 | 81
  Failure | 70 | 93
  Unknown/Missing (excluded from analysis) | 7 | 2
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Chi-squared test was used to calculate p-value. P-value was calculated for participants with clinical outcome as "cure"; Test type: Non-Inferiority or Equivalence — The final p-value was compared against an O'Brien-Fleming boundary of 0.048; p = 0.042, Chi-squared

2. Secondary Outcome: Clinical Outcome in Participants With Baseline MRSA at EOS for mITT Population
Description: as for outcome 1
Time Frame: EOS (7-30 days after last dose)
Population: mITT population included all ITT participants who received at least 1 dose of drug with a diagnosis of nosocomial pneumonia caused by proven MRSA and had an observed outcome for that visit unless already declared a failure prior to that visit.
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 186 | 205
Participants
  Cure | 102 | 92
  Failure | 84 | 113
  Unknown/Missing (excluded from analysis) | 38 | 19

3. Secondary Outcome: Clinical Outcome in Participants With Baseline MRSA at End of Treatment (EOT) for PP Population
Description: Clinical response evaluated at EOT visit as Cure:resolution of clinical sign/symptoms of pneumonia when compared with baseline;Improvement: in 2 or more clinical sign/symptoms of pneumonia when compared with baseline,improvement/lack of progression of all chest X-ray abnormalities,Failure: persistence/ progression of baseline signs/symptoms of pneumonia or baseline radiographic abnormalities after atleast 2 days of treatment; development of new pulmonary/extrapulmonary clinical findings consistent with active infection;Unknown: extenuating circumstances precluding classification to 1 of above.
Time Frame: EOT (within 72 hours of last dose)
Population: PP population included all mITT participants who satisfied all critical inclusion/exclusion criteria,had adequate dosing of drug (defined as 5 full days for success or 2 full days of treatment for participants whose clinical outcome was considered failure)and had observed outcome for that visit unless already declared failure prior to that visit.
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 180 | 186
Participants
  Cure | 76 | 70
  Improvement | 74 | 60
  Failure | 30 | 56
  Unknown/Missing (excluded from analysis) | 3 | 2

4. Secondary Outcome: Clinical Outcome in Participants With Baseline MRSA at EOT for mITT Population
Description: as for outcome 3
Time Frame: EOT (within 72 hours of last dose)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 201 | 214
Participants
  Cure | 81 | 77
  Improvement | 80 | 68
  Failure | 40 | 69
  Unknown/Missing (excluded from analysis) | 23 | 10

5. Secondary Outcome: Microbiological Outcome in Participants With Baseline MRSA at EOS for PP Population
Description: Microbiological response assessed at participant level.Eradication:baseline isolate not present in repeat culture from original infection site;Presumed Eradication:clinical response of cure precluded availability of specimen for culture;Persistence:baseline isolate present in repeat culture;Presumed Persistence:culture data not available for participant with clinical response of failure;Superinfection:culture from primary infection site had new pathogen not identified as baseline isolate and clinical response was failure;Indeterminate:any participant who cannot be classified into any of above.
Time Frame: EOS (7-30 days after last dose)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 167 | 174
Participants
  MRSA Eradication | 35 | 26
  Presumed MRSA Eradication | 62 | 56
  MRSA Persistence | 7 | 15
  MRSA Recurrence | 15 | 11
  Presumed MRSA Persistence | 48 | 66
  Missing/Indeterminate (excluded from analysis) | 5 | 2

6. Secondary Outcome: Microbiological Outcome in Participants With Baseline MRSA at EOS for mITT Population
Description: as for outcome 5
Time Frame: EOS (7-30 days after last dose)
Population: mITT population included all ITT participants (who received at least 1 dose of drug) with a diagnosis of nosocomial pneumonia caused by proven MRSA and had an observed outcome for that visit unless already declared a failure prior to that visit.
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 195 | 209
Participants
  MRSA Eradication | 46 | 35
  Presumed MRSA Eradication | 65 | 61
  MRSA Persistence | 9 | 22
  MRSA Recurrence | 16 | 12
  Presumed MRSA Persistence | 59 | 79
  Missing/Indeterminate (excluded from analysis) | 29 | 15

7. Secondary Outcome: Microbiological Outcome in Participants With Baseline MRSA at EOT for PP Population
Description: as for outcome 5
Time Frame: EOT (within 72 hours of last dose)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 182 | 188
Participants
  MRSA Eradication | 76 | 59
  Presumed MRSA Eradication | 73 | 55
  MRSA Persistence | 16 | 50
  Presumed MRSA Persistence | 17 | 24
  Missing/Indeterminate (excluded from analysis) | 1 | 0

8. Secondary Outcome: Microbiological Outcome in Participants With Baseline MRSA at EOT for mITT Population
Description: as for outcome 5
Time Frame: EOT (within 72 hours of last dose)
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 203 | 218
Participants
  MRSA Eradication | 84 | 65
  Presumed MRSA Eradication | 77 | 62
  MRSA Persistence | 19 | 60
  Presumed MRSA Persistence | 23 | 31
  Missing/Indeterminate (excluded from analysis) | 21 | 6

9. Secondary Outcome: Number of Participants With Clinical Signs and Symptoms at EOS for PP Population
Description: Participant's clinical evaluation of signs and symptoms were based on global assessment by investigator at specific timepoints. Signs and symptoms (mild to severe) of nosocomial pneumonia included cough; production of purulent sputum or change in character of sputum;auscultatory findings on pulmonary examination of rales and/or pulmonary consolidation (dullness on percussion, bronchial breath sounds, or egophony); and dyspnea, tachypnea, or hypoxemia with PaO2 <60 mmHg or worsening gas exchange or increased oxygen requirements; pleuritic chest pain; chills/rigors; and decreased breath sounds.
Time Frame: EOS (7-30 days after last dose)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 172 | 176
Participants
  Decreased Breath Sounds | 42 | 46
  Hypoxia | 30 | 29
  Pulmonary Consolidation | 22 | 19
  Rales | 27 | 27
  Tachypnea | 39 | 36
  Chills/Rigors | 3 | 1
  Cough | 32 | 33
  Dyspnea | 15 | 19
  Pleuritic Chest Pain | 5 | 5
  Purulent Sputum | 36 | 26

10. Secondary Outcome: Number of Participants With Clinical Signs and Symptoms at EOS for mITT Population
Description: as for outcome 9
Time Frame: EOS (7-30 days after last dose)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 224 | 224
Participants
  Decreased Breath Sounds | 53 | 58
  Hypoxia | 38 | 38
  Pulmonary Consolidation | 32 | 27
  Rales | 36 | 34
  Tachypnea | 49 | 42
  Chills/Rigors | 4 | 2
  Cough | 37 | 40
  Dyspnea | 19 | 23
  Pleuritic Chest Pain | 7 | 6
  Purulent Sputum | 48 | 38

11. Secondary Outcome: Number of Participants With Clinical Signs and Symptoms at EOT for PP Population
Description: as for outcome 9
Time Frame: EOT (within 72 hours of last dose)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 183 | 188
Participants
  Decreased Breath Sounds | 63 | 99
  Hypoxia | 56 | 60
  Pulmonary Consolidation | 43 | 69
  Rales | 49 | 61
  Tachypnea | 67 | 58
  Chills/Rigors | 3 | 0
  Cough | 53 | 59
  Dyspnea | 24 | 27
  Pleuritic Chest Pain | 2 | 1
  Purulent Sputum | 55 | 74

12. Secondary Outcome: Number of Participants With Clinical Signs and Symptoms at EOT for mITT Population
Description: as for outcome 9
Time Frame: EOT (within 72 hours of last dose)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 224 | 224
Participants
  Decreased Breath Sounds | 73 | 109
  Hypoxia | 67 | 73
  Pulmonary Consolidation | 53 | 77
  Rales | 57 | 73
  Tachypnea | 76 | 66
  Chills/Rigors | 5 | 2
  Cough | 64 | 64
  Dyspnea | 28 | 33
  Pleuritic Chest Pain | 4 | 2
  Purulent Sputum | 67 | 85

13. Secondary Outcome: Survival Status Estimated by Kaplan-Meier Analysis for PP Population
Description: For each participant, time to death was estimated from baseline to date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 days after last dose. The distribution of survival was estimated for the treatment groups using the Kaplan-Meier, product-limit method and compared between the treatment groups using the log rank statistic.
Time Frame: From baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 days after last dose.
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 183 | 188
Days | 59.196 (1.684) | 57.191 (1.686)
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Statistical comparison of survival analysis was performed.Log rank method was used to calculate p-value; Test type: Superiority or Other; p = 0.9344, Log Rank

14. Secondary Outcome: Survival Status Estimated by Kaplan-Meier Analysis for mITT Population
Description: as for outcome 13
Time Frame: as for outcome 13
Population: mITT population included all ITT participants (who received at least 1 dose of drug) with a diagnosis of nosocomial pneumonia caused by proven MRSA.
Measure: Median (Standard Error); unit: Days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 224 | 224
Days | 58.185 (1.605) | 57.072 (1.570)
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Statistical comparison of survival analysis was performed.Log rank method was used to calculate p-value; Test type: Superiority or Other; p = 0.5985, Log Rank

15. Secondary Outcome: Survival Status Estimated by Kaplan-Meier Analysis for ITT Population
Description: as for outcome 13
Time Frame: as for outcome 13
Population: ITT population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 597 | 587
Days | 55.590 (1.511) | 55.369 (1.484)
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Statistical comparison of survival analysis was performed.Log rank method was used to calculate p-value; Test type: Superiority or Other; p = 0.8590, Log Rank

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Linezolid | Vancomycin
Serious Adverse Events (participants affected / at risk) | 145/597 | 141/587
Other Adverse Events (participants affected / at risk) | 348/597 | 381/587
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linezolid (N=597) | Vancomycin (N=587)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 3
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 11 | 13
Cardiac failure congestive (Cardiac disorders) | 1 | 5
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 9 | 4
Cardiogenic shock (Cardiac disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Electromechanical dissociation (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal dilatation (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 2
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Drug ineffective (General disorders) | 1 | 0
Multi-organ disorder (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 7 | 3
Pyrexia (General disorders) | 2 | 0
Secretion discharge (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Abdominal sepsis (Infections and infestations) | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 1
Acinetobacter bacteraemia (Infections and infestations) | 0 | 1
Acinetobacter infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 1
Candidiasis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 1
Clostridium colitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Fungal sepsis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 2
Meningitis bacterial (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 14 | 9
Pneumonia bacterial (Infections and infestations) | 1 | 3
Pneumonia klebsiella (Infections and infestations) | 2 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 3
Post procedural sepsis (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Pyothorax (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 9 | 19
Septic shock (Infections and infestations) | 9 | 16
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 2 | 0
Systemic candida (Infections and infestations) | 1 | 2
Toxic shock syndrome streptococcal (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Anastomotic complication (Injury, poisoning and procedural complications) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0
Failure to anastomose (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteric cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain compression (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 3 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 3
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 2
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 2
Ischaemic stroke (Nervous system disorders) | 1 | 2
Mental impairment (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 0 | 1
Pneumocephalus (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Subdural hygroma (Nervous system disorders) | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 3
Azotaemia (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 6
Renal failure acute (Renal and urinary disorders) | 5 | 11
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 3 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dependence on respirator (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumon (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17 | 18
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Tracheal operation (Surgical and medical procedures) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Haemorrhage (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 5 | 6
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linezolid (N=597) | Vancomycin (N=587)
Anaemia (Blood and lymphatic system disorders) | 30 | 40
Coagulopathy (Blood and lymphatic system disorders) | 1 | 3
Eosinophilia (Blood and lymphatic system disorders) | 2 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 4 | 2
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 5
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 12
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 6
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 5 | 1
Arrhythmia (Cardiac disorders) | 4 | 2
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 10 | 13
Atrial flutter (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 9 | 7
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 3
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Cyanosis (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 7 | 5
Tachycardia (Cardiac disorders) | 11 | 11
Torsade de pointes (Cardiac disorders) | 1 | 0
Ventricular dysfunction (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 2 | 1
Ventricular tachycardia (Cardiac disorders) | 6 | 5
Ear pain (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 3 | 0
Diabetes insipidus (Endocrine disorders) | 1 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 2 | 6
Corneal disorder (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 2
Ocular discomfort (Eye disorders) | 0 | 1
Pupillary reflex impaired (Eye disorders) | 0 | 1
Pupils unequal (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 6 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Anal ulcer (Gastrointestinal disorders) | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 33 | 37
Diarrhoea (Gastrointestinal disorders) | 59 | 56
Dry mouth (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Dysphagia (Gastrointestinal disorders) | 7 | 8
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastric hypomotility (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 4
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 2
Ileus (Gastrointestinal disorders) | 5 | 3
Ileus paralytic (Gastrointestinal disorders) | 3 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 22 | 29
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Perianal erythema (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Tooth loss (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 14 | 14
Asthenia (General disorders) | 1 | 4
Catheter site erythema (General disorders) | 0 | 1
Catheter site haematoma (General disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 1 | 1
Catheter site pain (General disorders) | 0 | 3
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 3
Device malfunction (General disorders) | 0 | 1
Device occlusion (General disorders) | 3 | 5
Face oedema (General disorders) | 0 | 1
Generalised oedema (General disorders) | 11 | 4
Hyperthermia (General disorders) | 2 | 0
Hypothermia (General disorders) | 0 | 6
Implant site effusion (General disorders) | 1 | 0
Infusion site erythema (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 2
Infusion site oedema (General disorders) | 1 | 0
Infusion site phlebitis (General disorders) | 3 | 5
Infusion site swelling (General disorders) | 0 | 1
Infusion site thrombosis (General disorders) | 2 | 0
Irritability (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 2
Medical device complication (General disorders) | 1 | 0
Medical device pain (General disorders) | 1 | 1
Multi-organ disorder (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema (General disorders) | 3 | 2
Oedema peripheral (General disorders) | 12 | 13
Pain (General disorders) | 10 | 5
Puncture site haemorrhage (General disorders) | 0 | 1
Pyrexia (General disorders) | 22 | 24
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Thrombosis in device (General disorders) | 1 | 1
Vessel puncture site haematoma (General disorders) | 0 | 1
Vessel puncture site pain (General disorders) | 1 | 0
Xerosis (General disorders) | 1 | 0
Biliary fistula (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholestasis (Hepatobiliary disorders) | 2 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2
Jaundice (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 1 | 0
Acinetobacter infection (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 4 | 4
Bacterial disease carrier (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Bacteriuria (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 1
Candida sepsis (Infections and infestations) | 1 | 1
Candidiasis (Infections and infestations) | 4 | 5
Candiduria (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 3
Cellulitis (Infections and infestations) | 4 | 2
Citrobacter infection (Infections and infestations) | 2 | 0
Clostridial infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 7 | 6
Conjunctivitis bacterial (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 3 | 2
Device related sepsis (Infections and infestations) | 0 | 2
Enterobacter bacteraemia (Infections and infestations) | 1 | 0
Enterobacter pneumonia (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 2 | 0
Fungal cystitis (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 6 | 5
Fungal sepsis (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 6 | 8
Gastrointestinal infection (Infections and infestations) | 1 | 0
Genital infection fungal (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infectious disease carrier (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 0 | 1
Infusion site cellulitis (Infections and infestations) | 1 | 0
Infusion site infection (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 1 | 2
Lung abscess (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 5 | 0
Lung infection pseudomonal (Infections and infestations) | 6 | 4
Mastitis fungal (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 6 | 5
Oral fungal infection (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 1 | 3
Osteomyelitis (Infections and infestations) | 1 | 0
Pancreatic abscess (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1
Pleural infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 11
Pneumonia bacterial (Infections and infestations) | 4 | 5
Pneumonia escherichia (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 2 | 3
Pneumonia staphylococcal (Infections and infestations) | 1 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 3
Postoperative wound infection (Infections and infestations) | 3 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 3
Rash pustular (Infections and infestations) | 0 | 1
Respiratory moniliasis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 1 | 3
Sinusitis (Infections and infestations) | 1 | 1
Skin candida (Infections and infestations) | 1 | 4
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1
Stenotrophomonas infection (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 1
Tracheitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 2 | 2
Tracheostomy infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 29 | 19
Urinary tract infection fungal (Infections and infestations) | 3 | 5
Urinary tract infection pseudomonal (Infections and infestations) | 3 | 2
Vulvovaginal candidiasis (Infections and infestations) | 2 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 0 | 2
Wound infection bacterial (Infections and infestations) | 1 | 0
Wound infection fungal (Infections and infestations) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Anal injury (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 2
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 2
Eschar (Injury, poisoning and procedural complications) | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 3 | 5
Fall (Injury, poisoning and procedural complications) | 1 | 1
Feeding tube complication (Injury, poisoning and procedural complications) | 2 | 1
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 1 | 2
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 0 | 1
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 2
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 2 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 6
Post procedural oedema (Injury, poisoning and procedural complications) | 2 | 2
Post-thoracotomy pain syndrome (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 6 | 5
Pulmonary radiation injury (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 5 | 4
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Acid base balance abnormal (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 3
Antibiotic resistant Staphylococcus test positive (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 3
Bacterial test positive (Investigations) | 2 | 4
Blood albumin decreased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 1
Blood amylase increased (Investigations) | 1 | 4
Blood bicarbonate decreased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 3 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood chloride decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 4
Blood culture positive (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 4 | 4
Blood magnesium decreased (Investigations) | 0 | 2
Blood phosphorus decreased (Investigations) | 1 | 2
Blood potassium decreased (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 1 | 1
Blood pressure increased (Investigations) | 3 | 3
Blood sodium decreased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Carbon dioxide increased (Investigations) | 0 | 1
Cardiac enzymes increased (Investigations) | 0 | 1
Chest X-ray abnormal (Investigations) | 0 | 1
Clostridium test (Investigations) | 1 | 0
Coagulation time prolonged (Investigations) | 0 | 1
Fungal test positive (Investigations) | 4 | 2
Gastric occult blood positive (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 2 | 3
Heart rate increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 3 | 5
Lipase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 4 | 1
Neutrophil count increased (Investigations) | 1 | 0
Occult blood positive (Investigations) | 2 | 1
Oxygen saturation decreased (Investigations) | 1 | 2
Pedal pulse decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 2 | 0
Platelet count increased (Investigations) | 4 | 1
Prothrombin level decreased (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 2
Pulse abnormal (Investigations) | 0 | 1
Radial pulse decreased (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 1 | 0
Reticulocyte count increased (Investigations) | 1 | 1
Spirometry abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 3 | 5
Troponin increased (Investigations) | 2 | 0
Urine output decreased (Investigations) | 0 | 2
Urine sodium increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 0
White blood cell count increased (Investigations) | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Cell death (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Electrolyte depletion (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 6
Fluid overload (Metabolism and nutrition disorders) | 10 | 11
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 18
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 12
Hyperlactacidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 3
Hypernatraemia (Metabolism and nutrition disorders) | 7 | 8
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | 7
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 21 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 44 | 43
Hypomagnesaemia (Metabolism and nutrition disorders) | 16 | 15
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 13
Hypophosphataemia (Metabolism and nutrition disorders) | 11 | 11
Hypovolaemia (Metabolism and nutrition disorders) | 3 | 1
Iron overload (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 4 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 4 | 4
Metabolic alkalosis (Metabolism and nutrition disorders) | 6 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Aphonia (Nervous system disorders) | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 3 | 3
Convulsions local (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 8
Hemiparesis (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 2
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 3
Mental impairment (Nervous system disorders) | 2 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 1
Muscle spasticity (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Neuromuscular blockade (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Paralysis flaccid (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 2 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1
Radial nerve palsy (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 3 | 1
Syncope (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 3
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Affective disorder (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 13 | 22
Anxiety (Psychiatric disorders) | 11 | 15
Confusional state (Psychiatric disorders) | 5 | 1
Delirium (Psychiatric disorders) | 4 | 2
Depression (Psychiatric disorders) | 12 | 7
Disorientation (Psychiatric disorders) | 3 | 0
Hallucination (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 14 | 18
Mental status changes (Psychiatric disorders) | 1 | 3
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 2 | 2
Restlessness (Psychiatric disorders) | 5 | 3
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 5
Chromaturia (Renal and urinary disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 3 | 4
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 6 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Pyuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 8
Renal failure acute (Renal and urinary disorders) | 5 | 9
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 3 | 3
Urethral pain (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 3 | 1
Genital rash (Reproductive system and breast disorders) | 2 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 1
Penile discharge (Reproductive system and breast disorders) | 1 | 0
Penile swelling (Reproductive system and breast disorders) | 0 | 1
Prostatism (Reproductive system and breast disorders) | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 1 | 3
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dependence on respirator (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurocutaneous fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pneumothorax spontaneous tension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Blister (Skin and subcutaneous tissue disorders) | 2 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 16 | 23
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 4
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Plantar erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 22 | 20
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papulosquamous (Skin and subcutaneous tissue disorders) | 1 | 0
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 4 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 2
Skin maceration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 | 4
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 6
Flushing (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hyperaemia (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 28 | 33
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 21 | 35
Phlebitis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 2 | 0
Influenza virus test positive (Investigations) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Embolism arterial (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
EOS visit window of 15-21 days after last dose as specified in protocol was expanded during blinded evaluability assessments and prior to database lock and unblinding to 7-30 days after last dose in order to better fit the actual study visit days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.